CLINICAL TRIAL: NCT04297267
Title: A Prospective, Single Arm, Multicenter, Phase II Trial of Gemcitabine Plus Cisplatin in the Treatment of Patients With Non-pCR Triple Negative Breast Cancer Following Neoadjuvant Chemotherapy
Brief Title: A Study to Evaluate Gemcitabine Plus Cisplatin in the Treatment of TNBC Patients Following Neoadjuvant Chemotherapy
Acronym: nonpCR GP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608162-19-1805B
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Triple Negative Breast Cancer
Keywords: gemcitabine; cisplatin; non-pCR; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP group (Experimental): Patients should receive four cycles of GP regimen (cisplatin at 75 mg/m2 iv infusion on day 1 plus gemcitabine at 1250 mg/m2 iv infusion over 30 min on day 1 and 8 every 3 weeks).
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1250mg/m2,d1,d8,every 3 weeks
Drug: Cisplatin — Cisplatin 75mg/m2,d1，every 3 weeks

SUMMARY:
This is a prospective, open-lable phase II clinical trial evaluating the effectiveness and safety of gemcitabine plus cisplatin as adjuvant treatment for non-pCR TNBC patients after standard neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, open-lable phase II clinical trial evaluating the effectiveness and safety of gemcitabine plus cisplatin as adjuvant treatment for non-pCR TNBC patients after standard neoadjuvant chemotherapy. Non-pCR TNBC patients who completed 6-8 cycles of standard neoadjuvant chemotherapy will be included in this study and receive 4 cycles of GP regimen chemotherapy(cisplatin 75 mg/m² d1 and gemcitabine 1250 mg/m² d1,8, every 3 weeks). Our primary endpoint is disease free survival (DFS). Secondary end points include overall survival (OS), recurrence free survival (RFS), distant disease free survival (DDFS)rates and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Patients with histologically confirmed unilateral invasive ductal carcinoma(according to WHO histologically type)
* Tumor clinical staged as IIB-IIIB before neoadjuvant chemotherapy (according to the 7th AJCC edition).
* After standard treatment (6-8 cycles) of neoadjuvant chemotherapy (plan formulated by the attending doctor, including anthracycline and paclitaxel drugs, must not contain platinum), assessed by the surgery, the original site for non - pCR (MP class 1-4) or lymph nodes are still positive for patients.
* No gross or microscopic tumor residual after resection.
* Patients with clear ER/PR/Her2 receptor, and ER/PR/Her2 are all negative(Specific definition: immunohistochemical detection of ER < 1% positive tumor cell is defined as the ER negative, PR < 1% positive tumor cells is defined as the PR negative, Her2 0-1 or Her2 2 + but after FISH or CISH tested negatie for c (no amplification) is defined as the Her2-negative).
* No evidence of distant metastasis in the clinical or radiological aspects of preoperative. examination,that is M0.
* Patients without peripheral neuropathy or I peripheral neurotoxicity.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
* Patients recovered well after surgery, at least 1 weeks after the operation.
* Adequate marrow: White blood cells count≥3000/μL,neutrophil count ≥1500/μL, hemoglobin ≥9g/dL and platelet count ≥75000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ 1.5ULN.
* Adequate renal function: Serum creatinine ≤ 1.5ULN.
* Contraception during the treatment of child-bearing women.
* Adequate cardiac function :Left ventricular ejection fraction (LVEF) > 50%.
* Patients must be informed of the investigational nature of this study and give written informed consent.
* Patients without serious heart, lung, liver, kidney and other important organs disease history.
* Patients have good compliance.

Exclusion Criteria:

* Patients with bilateral breast cancer or carcinoma in situ(DCIS/LCIS).
* Metastasis of any part except axillary lymph nodes.
* Clinical or imaging suspicion of the contralateral breast is malignant but not confirmed, requiring biopsy.
* There have been malignant tumors (except for basal cell carcinoma and carcinoma in situ of cervix) in the last five years, including breast cancer.
* Patients have been enrolled in other clinical trials.
* Patients with severe systemic illnesses and/or uncontrolled infections are unable to join the study.
* Patients with severe cardio-cerebrovascular disorders (e.g., unstable angina pectoris, chronic heart failure, uncontrollable hypertension >160/100mmgh, myocardial infarction or cerebrovascular accident) in the first 6 months of randomization.
* Pregnant lactating women (child-bearing women must be negative for pregnancy test within 14 days prior to first delivery, if positive, the pregnancy should be excluded by ultrasound.)
* Child-bearing women who are unwilling to take effective contraceptive measures in the course of research.
* Patients with mental illness, cognitive impairment, inability to understand test protocols and side effects, and those who fail to complete the trial programme and follow-up work (a systematic assessment is required before the trial).
* Persons without personal freedom and independent civil capacity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3-year
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer

SECONDARY OUTCOMES:
Recurrence free survival | 3-year
  Recurrence free survival is calculated from surgery to the first recurrence.
Distant disease free survival | 3-year
  Distant disease free survival is calculated from surgery to the first distant metastasis.
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Disease free survival(5year) | 5-year
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer
Recurrence free survival(5year) | 5-year
  Recurrence free survival(5y) is calculated from surgery to the first recurrence.
Distant disease free survival(5year) | 5-year
  Distant disease free survival is calculated from surgery to the first distant metastasis.
Overall survival(5year) | 5-year
  Overall survival is calculated from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China